CLINICAL TRIAL: NCT03354884
Title: caBozantinib in cOllectiNg ductS Renal Cell cArcInoma (BONSAI)
Brief Title: caBozantinib in cOllectiNg ductS Renal Cell cArcInoma
Acronym: BONSAI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 150/17
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Collecting Duct Carcinoma (Kidney)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): All subjects will receive open label Cabozantinib 60 mg orally once daily
  Interventions: Drug: cabozantinib

INTERVENTIONS:
Drug: cabozantinib — cabozantinib 60 mg orally once daily

SUMMARY:
This is a single-arm, phase II trial (monocentric) study designed to determine To evaluate activity of Cabozantinib in terms of ORR according to the RECIST 1.1 criteria in Metastatic Collecting Duct Renal Cell Carcinoma

DETAILED DESCRIPTION:
This is a single-arm, phase II trial (monocentric)

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent Form
2. Unresectable, advanced or metastatic collecting ducts carcinoma untreated with any systemic agent for advanced disease
3. Measurable disease as defined by RECIST v1.1 criteria
4. Age ≥18 years
5. ECOG Performance Status 0-1
6. Any of the following laboratory test findings:

   * Hemoglobin > 9 g/dL (5.6 mmol/L)
   * WBC > 2,000/mm3
   * Neutrophils > 1,500/mm3
   * Platelets > 100,000/mm3
   * AST or ALT < 3 x ULN (< 5 x ULN if liver metastases are present)
   * Total Bilirubin < 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
   * Serum creatinine < 1.5 x upper limit of normal (ULN) or creatinine clearance ≥ 40 mL/min (measured or calculated by Cockroft-Gault formula)
   * Lipase < 2.0 x the upper limit of normal and no radiologic or clinical evidence of pancreatitis
   * PT-INR/PTT ≤ 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.] For patients on warfarin, close monitoring of at least weekly evaluations will be performed, until INR is stable based on a measurement at pre-dose, as defined by the local standard of care
7. Availability of a representative FFPE tumor specimen collected within 24 months of starting first-line cabozantinib that enables the definitive diagnosis of CDC (the archival specimen must contain adequate viable tumor tissue to enable candidate biomarkers status; the specimen may consist of a tissue block or at least 15 unstained serial sections; for core needle biopsy specimens, at least two cores should be available for evaluation)
8. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the study and for 4 months after the last dose of study treatment
9. Female subjects of childbearing potential must not be pregnant at screening

Exclusion Criteria:

1. Previous therapy for advanced disease; any medical adjuvant treatment must have been stopped at least six months before entry into the study
2. History of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
3. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].
4. History of cerebrovascular accidents, including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
5. Major surgery or trauma within 28 days before to study entry; the such as catheter placement not considered to be major surgery).
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before randomization.
7. Evidence of active bleeding or bleeding diathesis and/or clinically-significant GI bleeding within 6 months before the first dose of study treatment; 3 months for pulmonary hemorrhage and patients with tumor invading or encasing any major blood vessels.
8. Patients with GI disorders associated with a high risk of perforation or fistula formation.
9. Subjects with clinically relevant ongoing complications from prior radiation therapy.
10. Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
11. Previous or ongoing treatment (except for adjuvant therapies) with any of the following anti-cancer therapies: chemotherapy, immunotherapy, target therapies, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of Cabozantinib
12. Inability to swallow tablets or capsules.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 30 Month
  To evaluate activity of Cabozantinib in terms of ORR according to the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression free Survival (PFS) | 30 Month
  To evaluate activity of Cabozantinib in terms of PFS
Overall survival (OS) | 30 Month
  To evaluate activity of Cabozantinib in terms of OS
Safety and Tolerability (Adverse Events) | 30 Month
  To evaluate tolerability of Cabozantinibv during the treatment in particular the Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori - Milano
Locations (1):
- Giuseppe Procopio, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbas M, Steffens S, Bellut M, Eggers H, Grosshennig A, Becker JU, Wegener G, Schrader AJ, Grunwald V, Ivanyi P. Intratumoral expression of programmed death ligand 1 (PD-L1) in patients with clear cell renal cell carcinoma (ccRCC). Med Oncol. 2016 Jul;33(7):80. doi: 10.1007/s12032-016-0794-0. Epub 2016 Jun 17. PMID 27317388
- [Background] Choueiri TK, Fay AP, Gray KP, Callea M, Ho TH, Albiges L, Bellmunt J, Song J, Carvo I, Lampron M, Stanton ML, Hodi FS, McDermott DF, Atkins MB, Freeman GJ, Hirsch MS, Signoretti S. PD-L1 expression in nonclear-cell renal cell carcinoma. Ann Oncol. 2014 Nov;25(11):2178-2184. doi: 10.1093/annonc/mdu445. Epub 2014 Sep 5. PMID 25193987
- [Background] Choueiri TK, Escudier B, Powles T, Mainwaring PN, Rini BI, Donskov F, Hammers H, Hutson TE, Lee JL, Peltola K, Roth BJ, Bjarnason GA, Geczi L, Keam B, Maroto P, Heng DY, Schmidinger M, Kantoff PW, Borgman-Hagey A, Hessel C, Scheffold C, Schwab GM, Tannir NM, Motzer RJ; METEOR Investigators. Cabozantinib versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1814-23. doi: 10.1056/NEJMoa1510016. Epub 2015 Sep 25. PMID 26406150
- [Background] Choueiri TK, Escudier B, Powles T, Tannir NM, Mainwaring PN, Rini BI, Hammers HJ, Donskov F, Roth BJ, Peltola K, Lee JL, Heng DYC, Schmidinger M, Agarwal N, Sternberg CN, McDermott DF, Aftab DT, Hessel C, Scheffold C, Schwab G, Hutson TE, Pal S, Motzer RJ; METEOR investigators. Cabozantinib versus everolimus in advanced renal cell carcinoma (METEOR): final results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2016 Jul;17(7):917-927. doi: 10.1016/S1470-2045(16)30107-3. Epub 2016 Jun 5. PMID 27279544
- [Background] Choueiri TK, Halabi S, Sanford BL, Hahn O, Michaelson MD, Walsh MK, Feldman DR, Olencki T, Picus J, Small EJ, Dakhil S, George DJ, Morris MJ. Cabozantinib Versus Sunitinib As Initial Targeted Therapy for Patients With Metastatic Renal Cell Carcinoma of Poor or Intermediate Risk: The Alliance A031203 CABOSUN Trial. J Clin Oncol. 2017 Feb 20;35(6):591-597. doi: 10.1200/JCO.2016.70.7398. Epub 2016 Nov 14. PMID 28199818
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Gabrilovich DI, Ostrand-Rosenberg S, Bronte V. Coordinated regulation of myeloid cells by tumours. Nat Rev Immunol. 2012 Mar 22;12(4):253-68. doi: 10.1038/nri3175. PMID 22437938
- [Background] Geissler K, Fornara P, Lautenschlager C, Holzhausen HJ, Seliger B, Riemann D. Immune signature of tumor infiltrating immune cells in renal cancer. Oncoimmunology. 2015 Feb 3;4(1):e985082. doi: 10.4161/2162402X.2014.985082. eCollection 2015 Jan. PMID 25949868
- [Background] Iacovelli R, Nole F, Verri E, Renne G, Paglino C, Santoni M, Cossu Rocca M, Giglione P, Aurilio G, Cullura D, Cascinu S, Porta C. Prognostic Role of PD-L1 Expression in Renal Cell Carcinoma. A Systematic Review and Meta-Analysis. Target Oncol. 2016 Apr;11(2):143-8. doi: 10.1007/s11523-015-0392-7. PMID 26429561
- [Background] Leite KR, Reis ST, Junior JP, Zerati M, Gomes Dde O, Camara-Lopes LH, Srougi M. PD-L1 expression in renal cell carcinoma clear cell type is related to unfavorable prognosis. Diagn Pathol. 2015 Oct 15;10:189. doi: 10.1186/s13000-015-0414-x. PMID 26470780
- [Background] Oudard S, Banu E, Vieillefond A, Fournier L, Priou F, Medioni J, Banu A, Duclos B, Rolland F, Escudier B, Arakelyan N, Culine S; GETUG (Groupe d'Etudes des Tumeurs Uro-Genitales). Prospective multicenter phase II study of gemcitabine plus platinum salt for metastatic collecting duct carcinoma: results of a GETUG (Groupe d'Etudes des Tumeurs Uro-Genitales) study. J Urol. 2007 May;177(5):1698-702. doi: 10.1016/j.juro.2007.01.063. PMID 17437788
- [Background] Pecuchet N, Bigot F, Gachet J, Massard C, Albiges L, Teghom C, Allory Y, Mejean A, Escudier B, Oudard S. Triple combination of bevacizumab, gemcitabine and platinum salt in metastatic collecting duct carcinoma. Ann Oncol. 2013 Dec;24(12):2963-7. doi: 10.1093/annonc/mdt423. Epub 2013 Nov 4. PMID 24190963
- [Background] Powles T, Eder JP, Fine GD, Braiteh FS, Loriot Y, Cruz C, Bellmunt J, Burris HA, Petrylak DP, Teng SL, Shen X, Boyd Z, Hegde PS, Chen DS, Vogelzang NJ. MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014 Nov 27;515(7528):558-62. doi: 10.1038/nature13904. PMID 25428503
- [Background] Procopio G, Testa I, Iacovelli R, Grassi P, Verzoni E, Garanzini E, Colecchia M, Torelli T, De Braud F. Treatment of collecting duct carcinoma: current status and future perspectives. Anticancer Res. 2014 Feb;34(2):1027-30. PMID 24511050
- [Background] Procopio G, Verzoni E, Iacovelli R, Colecchia M, Torelli T, Mariani L. Is there a role for targeted therapies in the collecting ducts of Bellini carcinoma? Efficacy data from a retrospective analysis of 7 cases. Clin Exp Nephrol. 2012 Jun;16(3):464-7. doi: 10.1007/s10157-012-0589-3. Epub 2012 Jan 26. PMID 22278601
- [Background] Selli C, Amorosi A, Vona G, Sestini R, Travaglini F, Bartoletti R, Orlando C. Retrospective evaluation of c-erbB-2 oncogene amplification using competitive PCR in collecting duct carcinoma of the kidney. J Urol. 1997 Jul;158(1):245-7. doi: 10.1097/00005392-199707000-00079. PMID 9186368
- [Background] Shin SJ, Jeon YK, Kim PJ, Cho YM, Koh J, Chung DH, Go H. Clinicopathologic Analysis of PD-L1 and PD-L2 Expression in Renal Cell Carcinoma: Association with Oncogenic Proteins Status. Ann Surg Oncol. 2016 Feb;23(2):694-702. doi: 10.1245/s10434-015-4903-7. PMID 26464193
- [Background] Taube JM, Klein A, Brahmer JR, Xu H, Pan X, Kim JH, Chen L, Pardoll DM, Topalian SL, Anders RA. Association of PD-1, PD-1 ligands, and other features of the tumor immune microenvironment with response to anti-PD-1 therapy. Clin Cancer Res. 2014 Oct 1;20(19):5064-74. doi: 10.1158/1078-0432.CCR-13-3271. Epub 2014 Apr 8. PMID 24714771
- [Background] Walter S, Weinschenk T, Stenzl A, Zdrojowy R, Pluzanska A, Szczylik C, Staehler M, Brugger W, Dietrich PY, Mendrzyk R, Hilf N, Schoor O, Fritsche J, Mahr A, Maurer D, Vass V, Trautwein C, Lewandrowski P, Flohr C, Pohla H, Stanczak JJ, Bronte V, Mandruzzato S, Biedermann T, Pawelec G, Derhovanessian E, Yamagishi H, Miki T, Hongo F, Takaha N, Hirakawa K, Tanaka H, Stevanovic S, Frisch J, Mayer-Mokler A, Kirner A, Rammensee HG, Reinhardt C, Singh-Jasuja H. Multipeptide immune response to cancer vaccine IMA901 after single-dose cyclophosphamide associates with longer patient survival. Nat Med. 2012 Aug;18(8):1254-61. doi: 10.1038/nm.2883. Epub 2012 Jul 29. PMID 22842478
- [Derived] Procopio G, Sepe P, Claps M, Buti S, Colecchia M, Giannatempo P, Guadalupi V, Mariani L, Lalli L, Fuca G, de Braud F, Verzoni E. Cabozantinib as First-line Treatment in Patients With Metastatic Collecting Duct Renal Cell Carcinoma: Results of the BONSAI Trial for the Italian Network for Research in Urologic-Oncology (Meet-URO 2 Study). JAMA Oncol. 2022 Jun 1;8(6):910-913. doi: 10.1001/jamaoncol.2022.0238. PMID 35420628